CLINICAL TRIAL: NCT03752073
Title: Comparison of Two Mechanical Methods of Outpatient Ripening of the Cervix
Acronym: CORC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling patients
Sponsor: Ochsner Health System (Other)
Collaborators: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000397
Record Dates: First submitted 2018-10-04; First posted 2018-11-23 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Induction of Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Trans-cervical cervical balloon (Experimental): 17 F non-latex Foley catheter will be placed and balloon filled with 30 cc of sterile normal saline.
  Interventions: Device: Trans-cervical cervical balloon
- Hygroscopic cervical dilators (Experimental): Dilapan-S hygroscopic dilators will be placed into the cervix at the level of the internal os.
  Interventions: Device: Hygroscopic cervical dilator

INTERVENTIONS:
Device: Trans-cervical cervical balloon — Insertion of Foley Catheter
  Arms: Trans-cervical cervical balloon
Device: Hygroscopic cervical dilator — Insertion of Dilapan-s
  Arms: Hygroscopic cervical dilators

SUMMARY:
This is a randomized prospective trial of two mechanical methods of pre-induction cervical ripening agents.

DETAILED DESCRIPTION:
Term, low risk patients requesting elective induction of labor who desire pre-induction cervical ripening at home will be randomized to receive an outpatient trans-cervical ripening balloon (17 F non-latex Foley catheter) or hygroscopic cervical dilator (Dilapan-S). Patients present to the hospital for their scheduled induction of labor approximately 12 hours later.

We hypothesize that the trans-cervical balloon and hygroscopic dilators will show equivalent efficacy in cervical ripening, but that pain scores and patient satisfaction will be better with the hygroscopic dilators.

ELIGIBILITY:
Inclusion Criteria:

* Women between 39 and 41 weeks gestational age who desire elective induction of labor, based on reliable estimated gestational age (defined as ultrasonography performed before 14 weeks 0 days, or a certain last menstrual period consistent with ultrasonography performed before 21 weeks 0 days).

Exclusion Criteria:

* 1. Risk factors for placental insufficiency or intra-partum complication such as intra-uterine growth restriction, hypertensive disease, diabetes requiring insulin therapy, multiple gestation, history of previous hysterotomy, cholestasis of pregnancy, placental abnormalities including low lying placenta (< 2 cm from cervical os), maternal cardiac disease, maternal pulmonary disease, known fetal anomaly, fetal demise, etc.
* 2. Simplified Bishop score must be <6 and cervical dilation <2 cm.
* 3. Women must be able to give informed consent.
* 4. Concern regarding fetal well-being, conditions which preclude vaginal birth, group B strep carriers, patients who are HIV, Hep B or Hep C positive.
* 5. Women allergic to povidone-iodine, aquacryl hydrogel or the latex-free Foley catheter.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Time from start of cervical ripening to delivery | 720-2160 minutes
  Time in minutes from placement of cervical ripening agent to delivery

SECONDARY OUTCOMES:
Pain of insertion | First hour
  Patient assessment of pain on insertion using pain analog scale
Pain over duration of cervical ripening | 12-14 hours
  Patient assessment of pain on admission using pain analog scale
Patient satisfaction with cervical ripening agent | 24-36 hours
  Patient survey postpartum day #1 regarding cervical ripening experience

OTHER OUTCOMES:
Rate of device expulsion prior to admission | 12-14 hours
  Number of patients reporting expulsion of the device prior to planned admission
Rate of onset of labor prior to planned admission | 12-14 hours
  Number of patients presenting in active labor prior to planned admission divided by all enrolled patients
Rate of cesarean delivery | 12-36 hours
  Number of patients requiring cesarean delivery divided by number of all enrolled patients
Rate of operative vaginal delivery | 12-36 hours
  Number of patients requiring operative vaginal delivery divided by number of all enrolled patients
Incidence of shoulder dystocia | 12-36 hours
  Number of patients diagnosed with shoulder dystocia divided by number of all enrolled patients
Incidence of intra-amniotic infection | 12-36 hours
  Number of patients diagnosed with intra-amniotic infection (maternal temperature >38C, maternal (>120) or fetal (>160) tachycardia) divided by number of all enrolled patients
Incidence of post-partum hemorrhage | 12-36 hours
  Number of patients diagnosed with post-partu hemorrhage (QBL >1000 ml) divided by number of all enrolled patients
10 minute Apgar score <7 | 12-36 hours
  Number of infants with 10 minute Apgar score <7 divided by number of all enrolled patients
Base excess >12 | 12-36 hours
  Number of infants with base excess >12 divided by number of all enrolled patients
Umbilical cord gas pH <7 | 12-36 hours
  Number of infants with umbilical cord gas <7 divided by number of all enrolled patients
Composite score of adverse neonatal outcomes | 12-72 hours
  Composite of perinatal adverse outcomes (the need for respiratory support within 72 hours after birth, Apgar score of 3 or less at 5 minutes, hypoxic-ischemic encephalopathy, seizure, infection (confirmed sepsis or pneumonia), aspiration syndrome, birth trauma (bone fracture, neurologic injury, or retinal hemorrhage), intracranial or subgaleal hemorrhage, or hypotension requiring vasopressor support)
Composite score of serious maternal morbidity or mortality | 12-72 hours
  Composite score of serious maternal morbidity (e.g. uterine rupture, admission to intensive care unit, septicemia), or death.

CONTACTS AND LOCATIONS:
Overall Officials: Brigid McCue, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - Ochsner Baptist Hospital, New Orleans, Louisiana
  - Brigid McCue, Bay Shore, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164
- [Background] Sciscione AC, Bedder CL, Hoffman MK, Ruhstaller K, Shlossman PA. The timing of adverse events with Foley catheter preinduction cervical ripening; implications for outpatient use. Am J Perinatol. 2014 Oct;31(9):781-6. doi: 10.1055/s-0033-1359718. Epub 2013 Dec 17. PMID 24347259
- [Background] Gilson GJ, Russell DJ, Izquierdo LA, Qualls CR, Curet LB. A prospective randomized evaluation of a hygroscopic cervical dilator, Dilapan, in the preinduction ripening of patients undergoing induction of labor. Am J Obstet Gynecol. 1996 Jul;175(1):145-9. doi: 10.1016/s0002-9378(96)70264-8. PMID 8694040
- [Background] Shindo R, Aoki S, Yonemoto N, Yamamoto Y, Kasai J, Kasai M, Miyagi E. Hygroscopic dilators vs balloon catheter ripening of the cervix for induction of labor in nulliparous women at term: Retrospective study. PLoS One. 2017 Dec 22;12(12):e0189665. doi: 10.1371/journal.pone.0189665. eCollection 2017. PMID 29272277
- [Result] Kuper SG, Jauk VC, George DM, Edwards RK, Szychowski JM, Mazzoni SE, Wang MJ, Files P, Tita AT, Subramaniam A, Harper LM. Outpatient Foley Catheter for Induction of Labor in Parous Women: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jul;132(1):94-101. doi: 10.1097/AOG.0000000000002678. PMID 29889751
- [Derived] Lu AMR, Lin B, Shahani D, Demertzis K, Muscat J, Zabel E, Olson P, Manayan O, Nonnamaker E, Fest J, McCue B. Randomized control trial comparing hygroscopic cervical dilators to cervical ripening balloon for outpatient cervical ripening. Am J Obstet Gynecol MFM. 2024 Apr;6(4):101318. doi: 10.1016/j.ajogmf.2024.101318. Epub 2024 Feb 28. PMID 38417552
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264